CLINICAL TRIAL: NCT01886235
Title: A Pilot Study of Feasibility of Performing Intravital Microscopy in Melanoma Patients
Brief Title: Intravital Microscopy for Identifying Tumor Vessels in Patients With Stage IA-IV Melanoma That is Being Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 231512; NCI-2013-01052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 231512 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2013-06-25 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Melanoma; Stage IA Skin Melanoma; Stage IB Skin Melanoma; Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnosis (intravital microscopy) (Experimental): Patients receive fluorescein sodium IV followed by intravital microscopic observation over 10-15 minutes during excision of the melanoma.
  Interventions: Procedure: Diagnostic Microscopy; Drug: Fluorescein Sodium Injection; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Diagnostic Microscopy — Undergo intravital microscopy
Drug: Fluorescein Sodium Injection — Given IV
  Other Names: Fluorescite
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot clinical trial studies intravital microscopy for identifying tumor vessels in patients with stage IA-IV melanoma that is being removed by surgery. New imaging procedures, such as intravital microscopy, may determine the extent of melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of performing intravital microscopy on accessible human melanoma tumors during their standard course of treatment (i.e., wide local excision). (Part I)

SECONDARY OBJECTIVES:

I. To determine the blood flow velocity of the tumor vessels and tissue penetration of fluorescein (fluorescein sodium) as a marker of tumor vessel permeability. (Part II)

OUTLINE:

Patients receive fluorescein sodium intravenously (IV) followed by intravital microscopic observation over 10-15 minutes during excision of the melanoma.

After completion of study treatment, patients are followed up at 3 weeks and then periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Have measurable disease in their skin by direct visualization (visible lesion typically > 0.5 cm in maximal diameter); to perform a microscopic observation, the lesion will have to be visible by the naked eye, lined-up visually, and be able to interface with the microscope objective; a melanoma lesion that is smaller than 0.5 cm in diameter would present several obstacles to obtaining a reliable microscopic observation in the operating room; therefore, a visible lesion, at a minimum of 0.5 cm in diameter, is proposed for this study
* Melanoma tumor that requires a wide local excision in the operating room; this may include any stage of melanoma from stage IA to stage IV that requires a wide excision in the operating room
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* To determine any sensitivity to fluorescein, subject must have a skin prick test preoperatively (at the time of the preoperative visit and after signed informed consent for entry into this clinical trial is given); a negative skin prick test to fluorescein is an inclusion criteria

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Melanoma deposit is deemed inaccessible to microscopic observation during the operative procedure (i.e., lesion is less than 0.5 cm or is not clearly visible to the naked eye)
* Renal dysfunction as defined as a glomerular filtration rate (GFR) < 70
* Any known allergy or prior reaction to fluorescein; also, a positive skin prick test to fluorescein is considered an exclusion criteria and the patient would not be eligible for entry into this study
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to undergo observational study (may also include preoperative testing results including electrocardiogram [EKG], chest x-ray, or pulmonary function tests that preclude a wide excision in the operating room)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09-04 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Skitzki, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnosis (Intravital Microscopy)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Intravital Microscopy on Accessible Human Melanoma Tumors During Standard Local Excision
Description: A successful intravital microscopic observation will include the ability to identify tumor vessels, measure tumor vessel diameters, determine vessel density per 10 x field and visualize fluorescein within the tumor vessels.
Time Frame: Up to 2 months
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
percentage of participants | 70 [39.4 to 90.7]

2. Secondary Outcome: "Percentage of Participants With Any Adverse Event
Description: Percentage of participants with any adverse event. Described using upper one-sided 95% Clopper Pearson confidence limits.
Time Frame: Up to 5 years
Population: All treated and eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
percentage of participants | 40 [9.6 to 70.4]

3. Secondary Outcome: Blood Flow Rates
Description: Sample tumor characteristics obtained from the intervention will be characterized using descriptive statistics (mean, medians) and 95% confidence intervals.
Time Frame: Up to 2 months
Population: All treated and evaluable patients. Only 7 patients had data available, one patient had an unobservable tumor and two patients the fluorscein never made it to the tumor.
Measure: Mean (95% Confidence Interval); unit: micrometers per second
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 7
micrometers per second | 270 [206 to 334]

4. Secondary Outcome: Complication Rate
Description: Number of participants with an event that would disrupt the standard surgical procedure or create an adverse event that would not be anticipated from the standard surgery.
Time Frame: Up to 5 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: Median Overall Survival
Description: Assessed using Kaplan Meier and Proportional Hazards methods. Collected through routine follow-up processes.
Time Frame: Up to 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
months | NA [13.9 to NA] — the median and upper confidence limit were not reached

6. Secondary Outcome: Median Progression Free Survival
Description: Assessed using Kaplan Meier and Proportional Hazards methods. Collected through routine follow-up processes.
Time Frame: Up to 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
months | NA [13.9 to NA] — The median and upper confidence limit were not reached.

7. Secondary Outcome: Percentage of Participants With Treatment Response
Description: Treatment response was based upon the presence of a recurrence of the melanoma at either primary or metastatic sites.
Time Frame: Up to 5 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 31]

8. Secondary Outcome: Tumor Vasculature
Description: as for outcome 3
Time Frame: Up to 2 months
Population: Stringent dosing requirements precluded assessment of tumor vasculature endpoints. These measurements will be addressed in future studies.
Arm/Group | Diagnosis (Intravital Microscopy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Diagnosis (Intravital Microscopy)
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnosis (Intravital Microscopy) (N=10)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnosis (Intravital Microscopy) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Skin infection (Infections and infestations) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood magnesium increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes